CLINICAL TRIAL: NCT00437476
Title: Pilot, Multicenter, Randomized Study on Lopinavir/Ritonavir-Monotherapy vs Lopinavir/Ritonavir Plus Selected Nucs, in HIV/HCV ARV-Naive Coinfected Patients With Chronic Hepatitis C or Compensated Cirrhosis, Starting Treatment With Ribavirin and Pegylated Interferon
Brief Title: Lopinavir/Ritonavir Monotherapy Versus Standard Highly Active Antiretroviral Therapy (HAART) in HIV/HCV Coinfected Antiretroviral (ARV) Naive Patients Starting Treatment With Anti-HCV Therapy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS San Raffaele (Other)
Collaborators: Abbott (Industry); Hoffmann-La Roche (Industry)
Responsible Party: adriano lazzarin, IRCCS San Raffaele
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Kamon 1
Record Dates: First submitted 2007-02-20; First posted 2007-02-21 (Estimated); Last update posted 2009-02-06 (Estimated); Status verified 2009-02

CONDITIONS: HIV Infections; Hepatitis C
Keywords: HIV/HCV; HIV and HCV coinfected patients; Treatment Naive
MeSH Terms: conditions — HIV Infections; Hepatitis C | interventions — Ribavirin

ARMS (2):
- A (Experimental): LPV/r + selected NRTIs for 26 weeks, followed by LPV/r monotherapy and anti HCV drugs for 48 weeks. All the patients will be followed-up for 24 weeks after the end of anti-HCV drugs for the evaluation of SVR.As anti-HCV drugs the patients will receive PEG-IFNa 2a 180 mcg/week + Ribavirin 1-1.2 g/day . At the end of week 12 of combined therapy, only patients who will reach an early virological response will continue anti-HCV drugs.
  Interventions: Drug: LPV/r; Drug: Nucleoside Reverse Transcriptase Inhibitors; Drug: PEG-IFNa 2a; Drug: Ribavirin
- B (Active Comparator): LPV/r+ selected NRTIs for 24 weeks, followed by the same HAART and anti-HCV drugs for 48 weeks. At the end of the co-treatment for HCV/HIV, each subject will be treated for HIV infection according to physician decision. All the patients will be followed-up for 24 weeks after the end of anti-HCV drugs for the evaluation of SVR.As anti-HCV drugs the patients will receive PEG-IFNa 2a 180 mcg/week + Ribavirin 1-1.2 g/day . At the end of week 12 of combined therapy, only patients who will reach an early virological response will continue anti-HCV drugs.
  Interventions: Drug: LPV/r; Drug: Nucleoside Reverse Transcriptase Inhibitors; Drug: PEG-IFNa 2a; Drug: Ribavirin

INTERVENTIONS:
Drug: LPV/r — Lopinavir/Ritonavir 200/50 mg 2 cpr BID monotherapy - 26 weeks (A) or 24 weeks (B)
Drug: Nucleoside Reverse Transcriptase Inhibitors — NRTIs for 26 weeks (A) or 24 weeks (B)
Drug: PEG-IFNa 2a — PEG-IFNa 2a 180 mcg/week (48 weeks)
Drug: Ribavirin — Ribavirin 1-1.2 g/day (48 weeks)

SUMMARY:
The purpose of this study is to evaluate if the combination of Lpv/r monotherapy and anti-HCV drugs does not match with additional toxicity induced by the association of HAART and Peg-IFN + ritonavir in patients naive for HIV and HCV.

Secondary objective is to assess if Lpv/r monotherapy during HCV-treatment is associated with HIV efficacy vs optimized HAART.

DETAILED DESCRIPTION:
This is a pilot, randomised, open label, controlled clinical trial. All eligible patients (CD4 count > 200 and no PI resistance)will receive 26 weeks induction HAART (LPV/r + selected NUCS). At the end of induction period (Phase I), all subjects with negative HIV-RNA from at least two months, Hb > 11 g/dL and CD4 count > 350 cells/mmc will be randomised (1:1), to receive LPV/r new tabs (200/50 mg, 2 cpr BID) monotherapy (arm A) or to continue the same HAART (arm B), associated to anti-HCV therapy for other 48 weeks (Phase II). The number of subjects to recruit will be 60 subjects to start the induction-phase with the aim to randomize, at least 25 subjects in each arm of the study. The total number of subjects to randomize will be 50. The Group A: will receive LPV/r + selected NRTIs for 26 weeks, followed by LPV/r monotherapy and anti HCV drugs for 48 weeks. Group B: will receive LPV/r+ selected NRTIs for 24 weeks, followed by the same HAART and anti-HCV drugs for 48 weeks. At the end of the co-treatment for HCV/HIV, each subject will be treated for HIV infection according to physician decision.All the patients will be followed-up for 24 weeks after the end of anti-HCV drugs for the evaluation of SVR.As anti-HCV drugs the patients will receive PEG-IFNa 2a 180 mcg/week + Ribavirin 1-1.2 g/day . At the end of week 12 of combined therapy, only patients who will reach an early virological response will continue anti-HCV drugs.

ELIGIBILITY:
Inclusion Criteria:

* Subject is >18 years old
* Subject has given written informed consent
* Serologic evidence of HIV infection by HIV antibody and HIV-RNA detection
* Serologic evidence of HCV infection by HCV antibody and HCV-RNA detection
* Subject is naive for HIV and HCV therapy
* Subject has active chronic hepatitis or compensated cirrhosis (Child-Pugh class A)
* Subject has a CD4+ count > 200 cell/mm3 and <500 cell/mm3.
* Subject has genotype available at baseline and no mutations (IAS)associated with resistance to antiretroviral drugs used.
* Subject and partner will use effective contraceptive methods for the duration of the study

Exclusion Criteria:

* Subject is HbsAg positive
* Subject has cirrhosis score Child-Pugh B/C, no previous hepatic decompensation
* Subject has HIV-related thrombocytopenia (Platelets count < 50.000 mmc)
* Subject has neutrophils count < 1500/mmc
* Subject has Hb value < 9 g/dL at screening and <11 g/dL at randomization
* Subject has creatinine value > 1.5 mg/dL
* Subject is on a HAART regimen included ddI and/or AZT
* Subject is pregnant or wishes to become so
* Subject has any cause of liver disease other than chronic hepatitis C, status of liver decompensation or any other condition consistent with decompensated liver disease (bleeding from esophageal varices, signs of current bleeding, significant ascites, hepatic encephalopathy)
* Subject is alcohol abuser (> 30 gr/die)
* Prior treatment with PEG-IFN/ribavirin
* Illicit drugs abuse that in the opinion of the investigator could lead to poor compliance with the terms of the protocol (maintenance treatment with methadone allowed)
* Active heart disease (e.g. angina, congestive heart failure, recent myocardial infarction, or significant arrhythmia)
* Subject has pre-existing severe depression, condition of severe psychiatric disorders such as suicidal ideation, suicide attempts, depression or acute psychosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-02; Primary Completion 2010-07 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
To assess if the combination of LPV/r monotherapy in association with | 18 months
anti-HCV therapy (PEG IFN alfa 2a + Ribavirin) does not match with additional | 18 months
toxicity induced by the combination of optimized HAART (Lopinavir/ritonavir + selected Nucs) and PEG-IFN alfa 2a+Ribavirin | 18 months
in patients naïve for HIV and HCV | 18 months

SECONDARY OUTCOMES:
To assess if LPV/r monotherapy during the HCV treatment | 18 and 24 months
is associated with anti HIV efficacy and a better patient satisfaction | 18 and 24 months
vs optimized HAART. | 18 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Adriano Lazzarin, MD, Principal Investigator — IRCCS San Raffaele Hospital
Locations (1):
- San Raffaele Hospital Dep. Infectious Diseases, Milan, Italy